CLINICAL TRIAL: NCT02245568
Title: An Open-Label, Extension Study of the Effects of LMTM in Subjects With Alzheimer's Disease or Behavioral Variant Frontotemporal Dementia (bvFTD)
Brief Title: Open-Label Study of Leuco-methylthioninium Bis(Hydromethanesulfonate) (LMTM) in Subjects With Alzheimer's Disease or Behavioral Variant Frontotemporal Dementia (bvFTD)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: This study has been terminated for administrative reasons only.
Sponsor: TauRx Therapeutics Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TRx-237-020
Expanded Access: NCT03539380 (Available)
Record Dates: First submitted 2014-08-27; First posted 2014-09-19 (Estimated); Results first posted 2020-06-02 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Alzheimer's Disease; Behavioral Variant Frontotemporal Dementia
Keywords: Dementia; Alzheimer Disease; bvFTD; Frontotemporal Dementia; Neurodegenerative Diseases; Brain Diseases; Cognitive Disorders
MeSH Terms: conditions — Alzheimer Disease; Dementia; Frontotemporal Dementia; Neurodegenerative Diseases; Brain Diseases; Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- LMTM (Experimental)
  Interventions: Drug: LMTM

INTERVENTIONS:
Drug: LMTM — The initial LMTM dose was 200 mg/day (one 100-mg tablet twice daily), except in subjects with bvFTD who were taking a reduced dose (i.e., 100 mg/day) upon entering this extension study. The dose could be increased (after at least 13 weeks of treatment) or decreased (at any time at or after 2 weeks of treatment) by the Investigator in 100-mg increments or decrements. The maximum allowable dose was 300 mg/day (or in those countries where limited by a Competent Authority or Ethics Committee, 200 mg/day).

SUMMARY:
The purpose of this study is to provide subjects who have completed participation in a Phase 2 or Phase 3 trial of LMTM continued access to therapy and to evaluate the long-term safety of LMTM.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with all cause dementia and probable Alzheimer's disease at enrollment and who completed participation in one of the following three TauRx studies (inclusive of the 4-week post-treatment follow-up visit): TRx-237-005, TRx-237-008, or TRx-237-015.
* Subjects with a diagnosis of probable bvFTD at enrollment and who completed participation in TauRx study TRx-237-007 through Visit 9 (Week 52).
* Females, if of child-bearing potential, must practice true abstinence or continue to use adequate contraception and agree to maintain this throughout the study
* Subject, and/or, in the case of reduced decision-making capacity, legally acceptable representative(s) consistent with national law and ethics approval is/are able to read, understand, and provide written informed consent
* Has an identified adult caregiver who is willing to provide written informed consent for his/her own participation; is able to read, understand, and speak the designated language at the study site; either lives with the subject or sees the subject for ≥1 hour/day ≥3 days/week; agrees to accompany the subject to each study visit; and is able to verify daily compliance with study drug
* Able to comply with the study procedures

Exclusion Criteria:

* History of swallowing difficulties
* Pregnant or breastfeeding
* Clinically significant laboratory, pulse co-oximetry, electrocardiogram, or imaging abnormality (in originating study) or emergent intercurrent illness that, in the judgment of the principal investigator, could result in the risk of participation outweighing the potential benefit
* Current participation in, or intent to enroll in, another clinical trial of a drug, biologic, device, or medical food
* In Germany, subjects mandated to reside in a continuous care or assisted living facility or those whose willingness to participate in the clinical trial may be unduly influenced

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 913 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (135):
- United States (57):
  - Xenoscience, Inc / 21st Century Neurology, Phoenix, Arizona
  - Southern California Research, LLC, Fountain Valley, California
  - Feldman, Robert MD, Laguna Hills, California
  - Collaborative Neuroscience Network, Long Beach, California
  - The Shankle Clinic, Newport Beach, California
  - Neuro-Therapeutics, Inc., Pasadena, California
  - Pacific Research Network, San Diego, California
  - San Francisco Clinical Research Center, San Francisco, California
  - Memory and Aging Centre, San Francisco, California
  - Schuster Medical Research Institute, Sherman Oaks, California
  - Mile High Research Center, Denver, Colorado
  - Institute for Neurodegenerative Disorders, New Haven, Connecticut
  - Yale University School of Medicine, New Haven, Connecticut
  - Coastal Connecticut Research, LLC, New London, Connecticut
  - JEM Research, Atlantis, Florida
  - Bradenton Research Center, Bradenton, Florida
  - Meridien Research, Brooksville, Florida
  - Brain Matters Research, Delray Beach, Florida
  - MD Clinical, Hallandale, Florida
  - Mayo Clinic, Jacksonville, Florida
  - CNS Healthcare, Inc, Jacksonville, Florida
  - Miami Research Associates, Miami, Florida
  - Compass Research, LLC, Orlando, Florida
  - The Roskamp Institute, Inc., Sarasota, Florida
  - Axiom Clinical Research of Florida, Tampa, Florida
  - University of South Florida, Tampa, Florida
  - Compass Research, LLC - North Clinic, The Villages, Florida
  - iResearch Atlanta, Decatur, Georgia
  - Neurostudies.net, Decatur, Georgia
  - Alexian Brothers Neurosciences Institute, Elk Grove Village, Illinois
  - Ruan Neurology Clinic and Research Center, Des Moines, Iowa
  - ActivMed Practices & Research, Methuen, Massachusetts
  - Mayo Clinic, Alzheimer's Disease Research Center, Rochester, Minnesota
  - Neurological Research Center - Hattiesburg Clinic, Hattiesburg, Mississippi
  - Millennium Psychiatric Associates, Creve Coeur, Missouri
  - Memory Enhancement Center of America, Inc, Eatontown, New Jersey
  - The Atlantic Neuroscience Institute, Springfield, New Jersey
  - Advanced Memory Research Institute of NJ PC, Toms River, New Jersey
  - Neurological Associates of Albany, P. C., Albany, New York
  - SPRI, Brooklyn, New York
  - Columbia University Taub Institute, New York, New York
  - Research Foundation for Mental Hygiene, Inc., Orangeburg, New York
  - UNC Department of Neurology, Physicians Office Building, Chapel Hill, North Carolina
  - Clinical Trials of America, Inc, Winston-Salem, North Carolina
  - Neurobehavioral Clinical Research, Canton, Ohio
  - University Hospitals Case Medical Center, Neurology Clinical Trials Unit, Cleveland, Ohio
  - Rivus Wellness and Research Institute, Oklahoma City, Oklahoma
  - The Clinical Trial Center, LLC, Jenkintown, Pennsylvania
  - Hospital of the University of Pennsylvania, Department of Neurology, Philadelphia, Pennsylvania
  - RI Hospital, Providence, Rhode Island
  - Neurology Clinic, P.C., Cordova, Tennessee
  - Clinical Neuroscience Solutions CNS Healthcare, Memphis, Tennessee
  - FutureSearch Trials of Neurology, Austin, Texas
  - Senior Adults Specialty Research, Inc., Austin, Texas
  - FutureSearch Trials of Dallas, LP, Dallas, Texas
  - University of Virginia Adult Neurology, Primary Care Center, Charlottesville, Virginia
  - Independent Psychiatric Consultants, Waukesha, Wisconsin
- Australia (9):
  - Frontotemporal Research Group, Camperdown, New South Wales
  - Division of Rehabilitation and Aged Care, Hornsby, New South Wales
  - Southern Neurology Pty Limited, Kogarah, New South Wales
  - Discipline of Psychiatry, University of Queensland, Herston, Queensland
  - Royal Adelaide Hospital Memory Trials Centre, Adelaide, South Australia
  - Box Hill Hospital, Box Hill, Victoria
  - Medical and Cognitive Research Unit, Austin Health Heidelberg Repatriation Hospital, Heidelberg West, Victoria
  - McCusker Alzheimer's Research Foundation Inc, Nedlands, Western Australia
  - Neurodegenerative Disorders Research Pty Ltd, Subiaco, Western Australia
- Belgium (3):
  - University Hospital Ghent Department of Neurology, Ghent
  - Jessa Hospital, Hasselt
  - GZA Sint-Augustinus, Wilrijk
- Canada (10):
  - Heritage Medical Research Clinic, Calgary, Alberta
  - Okanagan Clinical Trials, Kelowna, British Columbia
  - University of British Columbia Hospital, Clinic for Alzheimer Disease and Related Disorders, Vancouver, British Columbia
  - Vancouver Island Health Authority, Victoria, British Columbia
  - True North Clinical Research Halifax Inc, Halifax, Nova Scotia
  - True North Clinical Research Kentville Inc, Kentville, Nova Scotia
  - Geriatric Clinical Trials Group, St. Joseph's Health Care, Parkwood Hospital Site, London, Ontario
  - Toronto Memory Program, Toronto, Ontario
  - Jewish General Hospital, Montreal, Quebec
  - McGill Centre for Studies in Aging, Alzheimer Disease Research Unit, Verdun, Quebec
- Croatia (2):
  - University Hospital Centre Zagreb, Department of Neurology, Zagreb
  - University Psychiatric Hospital Vrapče, Zagreb
- Finland (2):
  - University of Eastern Finland, Brain Research Unit Mediteknia, Kuopio
  - Clinical Research Services Turku (CRST), Turku
- France (3):
  - Hôpitaux Civils de Colmar, Colmar, Cedex
  - Centre de Recherche Clinique, Toulouse
  - Hôpital de Charpennes, Villeurbanne
- Germany (2):
  - Charité, University Medicine Berlin, CBF, Neurology, Berlin
  - Arzeneimittelforschung Leipzig GmbH, Leipzig
- Malaysia (3):
  - University Kuala Lumpur Royal College of Medicine, Ipoh
  - Hospital Sultan Ismail, Johor Bahru
  - University Malaya Medical Centre, Kuala Lumpur
- Erasmus University Medical Center, Rotterdam, Netherlands
- Psychiatry Hospital "Dr. Gheorghe Preda", Department of Psychiatry III, Sibiu, Romania
- Russia (7):
  - Non-governmental Healthcare Institution "Central Clinical Hospital #6 of the JSC "Russian Railways", Moscow
  - Mental Health Research Center of the Russian Academy of Medical Sciences, Gerontopsychiatry department, Moscow
  - Mental Health Research Center of the Russian Academy of Medical Sciences, Moscow
  - City Clinical Hospital #34, City Scientific Practical Neurological Center, Novosibirsk
  - City Geriatric Medical and Social Center, Saint Petersburg
  - Saint Petersburg Psychoneurological Research Institute n. a. V.M. Bekhterev, Saint Petersburg
  - State Budgetary Healthcare Institution of Sverdlovsk region "Sverdlovsk Regional Clinical Psychiatric Hospital", Yekaterinburg
- Singapore (2):
  - National University Hospital (NUH), Singapore
  - National Neuroscience Institute (NNI), Singapore
- South Korea (5):
  - Dong-A University Hospital, Busan
  - Gachon University Gil Medical Center, Incheon
  - Samsung Medical Center, Seoul
  - Seoul National University Boramae Medical Center, Seoul
  - Seoul National University Hospital, Seoul
- Spain (4):
  - Fundació ACE, Barcelona
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Viamed Montecanal, Zaragoza
- Taiwan (5):
  - Chang Gung Memorial Hospital, Kaohsiung, Kaohsiung City
  - China Medical University Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Memorial Hospital, Linkou, Taoyuan District
- United Kingdom (19):
  - Grampian NHS, Royal Cornhill Hospital, Aberdeen
  - RICE - The Research Institute for the Care of Older People, Bath
  - Belfast Health and Social Care Trust (BHSCT), Belfast
  - The Barberry Centre, Birmingham
  - MAC Clinical Research Ltd, Blackpool
  - MAC Clinical Research Ltd, Cannock
  - Sussex Partnership NHS Foundation Trust, Cognitive Treatment and Research Unit, Crowborough
  - St Margaret's Hospital Mental Health Unit, Epping
  - Cognition Health Ltd, Guildford
  - MAC Clinical Research Ltd, Leeds
  - Cognition Health Ltd., London
  - Imperial College Healthcare NHS Trust - Charing Cross Hospital, London
  - Leonard Wolfson Experimental Neurology Centre, London
  - MAC Clinical Research Ltd, Manchester
  - Nuffield Department of Clinical Neurosciences, Oxford
  - Redwoods Centre, Shrewsbury
  - Wessex Neurological Centre, Southampton General Hospital, Southampton
  - Memory Assessment and Research Centre (MARC), Southampton
  - Kingshill Research Centre, Victoria Hospital, Swindon

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Subjects who completed a Phase 2 or 3 study of LMTM were eligible to enroll, pending their ability to meet the inclusion/exclusion criteria. A total of 913 subjects enrolled; however, data for 16 subjects in Spain were later excluded (GCP issues) and 1 UK subject was never dosed. Thus, 896 subjects are included in all analyses except disposition.
Groups:
- LMTM 100-300 mg/Day: The initial LMTM dose was 200 mg/day (one 100-mg tablet twice daily), except in subjects with bvFTD who were taking a reduced dose (i.e., 100 mg/day) upon entering this extension study. The dose could be increased (after at least 13 weeks of treatment) or decreased (at any time at or after 2 weeks of treatment) by the Investigator in 100-mg increments or decrements. The maximum allowable dose was 300 mg/day (or in those countries where limited by a Competent Authority or Ethics Committee, 200 mg/day).
Period: Overall Study
Arm/Group | LMTM 100-300 mg/Day
Started | 913
Completed | 60
Not Completed | 853
Not completed — Study terminated by Sponsor | 346
Not completed — Adverse Event | 144
Not completed — Lack of Efficacy | 98
Not completed — Withdrawal by Caregiver | 85
Not completed — Withdrawal by Subject | 77
Not completed — Withdrawal by Legal Representative | 31
Not completed — Missing (Site closure) | 16
Not completed — Physician Decision | 14
Not completed — Non-compliance with study drug | 11
Not completed — Death | 9
Not completed — Blue staining | 6
Not completed — Worsening dementia/caregiver withdrawal | 6
Not completed — Intolerance/dosing issues/interruption | 5
Not completed — Lost to Follow-up | 5

BASELINE CHARACTERISTICS:
Population: A total of 913 subjects were enrolled, however, data for 16 subjects in Spain were excluded for analysis purposes and 1 UK subject was enrolled but never dosed; thus, 896 subjects are included in these analyses.
Arm/Group | LMTM 100-300 mg/Day
Number analyzed (Participants) | 896
Age, Continuous [Mean (Full Range); unit: years] | 69.2 [39 to 89]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 478
  Male | 418
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 24
  Not Hispanic or Latino | 864
  Unknown or Not Reported | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 6
  Asian | 72
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 18
  White | 783
  More than one race | 2
  Unknown or Not Reported | 14
Region of Enrollment [Number; unit: participants]
  Singapore | 22
  United States | 459
  United Kingdom | 161
  Malaysia | 8
  Russia | 35
  Spain | 23
  Canada | 51
  South Korea | 13
  Netherlands | 2
  Belgium | 12
  Finland | 18
  Taiwan | 16
  Australia | 41
  France | 11
  Germany | 12
  Croatia | 11
  Romania | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Serious or Non-serious Adverse Events
Description: Study-emergent adverse events (including the onset of new adverse events or worsening of pre-existing adverse events) were recorded from the time of first dose in this study to the end of study participation. All laboratory test, vital sign, or electrocardiogram parameter abnormalities deemed clinically significant by the Investigator were to be reported as adverse events.
Time Frame: Up to 34 months
Population: The safety population was composed of participants dosed with 100-300 mg LMTM who were used for analysis. Safety was assessed over time by means of adverse event and concomitant medication recording; clinical laboratory tests; vital sign measurements and weight; 12-lead electrocardiograms; and targeted physical and neurological examinations.
Measure: Count of Participants; unit: Participants
Arm/Group | LMTM 100-300 mg/Day
Number analyzed (Participants) | 896
Participants | 734

ADVERSE EVENTS:
Time Frame: Up to 34 months
Description: Study-emergent adverse events (including the onset of new adverse events or worsening of pre-existing adverse events) were recorded from the time of first dose in this study to the end of study participation. All laboratory test, vital sign, or electrocardiogram parameter abnormalities deemed clinically significant by the Investigator were to be reported as adverse events.
Arm/Group | LMTM 100-300 mg/Day
All-Cause Mortality (participants affected / at risk) | 15/896
Serious Adverse Events (participants affected / at risk) | 146/896
Other Adverse Events (participants affected / at risk) | 717/896
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LMTM 100-300 mg/Day (N=896)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Haemolytic anaemia (Blood and lymphatic system disorders) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Atrial flutter (Cardiac disorders) | 2 (2)
Atrioventricular block (Cardiac disorders) | 1 (1)
Bradycardia (Cardiac disorders) | 2 (3)
Cardiac arrest (Cardiac disorders) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 2 (2)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1)
Sick sinus syndrome (Cardiac disorders) | 1 (1)
Hydrocele (Congenital, familial and genetic disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Colitis microscopic (Gastrointestinal disorders) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Duodenal ulcer perforation (Gastrointestinal disorders) | 1 (1)
Faecaloma (Gastrointestinal disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Large intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Chest pain (General disorders) | 4 (4)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 2 (2)
Hypersensitivity (Immune system disorders) | 1 (1)
Appendicitis (Infections and infestations) | 3 (3)
Bacterial pyelonephritis (Infections and infestations) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Cholecystitis infective (Infections and infestations) | 1 (1)
Clostridium difficile infection (Infections and infestations) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 6 (6)
Sepsis (Infections and infestations) | 4 (5)
Urinary tract infection (Infections and infestations) | 11 (11)
Urosepsis (Infections and infestations) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 1 (1)
Facial bones fracture (Injury, poisoning and procedural complications) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 9 (9)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 2 (2)
Hip fracture (Injury, poisoning and procedural complications) | 2 (2)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 1 (1)
Pelvic fracture (Injury, poisoning and procedural complications) | 1 (1)
Pulmonary contusion (Injury, poisoning and procedural complications) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1)
Blood glucose increased (Investigations) | 1 (1)
Liver function test abnormal (Investigations) | 1 (1)
Weight decreased (Investigations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 4 (4)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1)
Hypovolaemia (Metabolism and nutrition disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 2 (2)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 (1)
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Breast cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Tonsil cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Altered state of consciousness (Nervous system disorders) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 2 (2)
Coordination abnormal (Nervous system disorders) | 1 (1)
Dementia (Nervous system disorders) | 1 (1)
Dementia Alzheimer's type (Nervous system disorders) | 3 (3)
Grand mal convlusion (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 1 (1)
Lacunar infarction (Nervous system disorders) | 1 (1)
Loss of consciousness (Nervous system disorders) | 2 (2)
Migraine (Nervous system disorders) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1)
Seizure like phenomena (Nervous system disorders) | 1 (1)
Serotonin syndrome (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 6 (7)
Transient ischaemic attack (Nervous system disorders) | 4 (4)
Tremor (Nervous system disorders) | 1 (1)
VIIth nerve paralysis (Nervous system disorders) | 1 (1)
Abnormal behavior (Psychiatric disorders) | 1 (1)
Aggression (Psychiatric disorders) | 3 (3)
Agitation (Psychiatric disorders) | 4 (4)
Confusional state (Psychiatric disorders) | 1 (1)
Delirium (Psychiatric disorders) | 3 (3)
Hallucination, visual (Psychiatric disorders) | 1 (1)
Hypersexuality (Psychiatric disorders) | 1 (1)
Mental status changes (Psychiatric disorders) | 3 (4)
Staring (Psychiatric disorders) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 3 (3)
Suicidal attempt (Psychiatric disorders) | 1 (1)
Bladder mass (Renal and urinary disorders) | 1 (1)
Bladder prolapse (Renal and urinary disorders) | 1 (1)
Cystitis noninfective (Renal and urinary disorders) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 2 (2)
Nephropathy (Renal and urinary disorders) | 1 (1)
Renal failure, acute (Renal and urinary disorders) | 2 (2)
Renal impairment (Renal and urinary disorders) | 1 (1)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1)
Uterine prolapse (Reproductive system and breast disorders) | 2 (2)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Circulatory collapse (Vascular disorders) | 2 (3)
Deep vein thrombosis (Vascular disorders) | 1 (1)
Hypertensive crisis (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 2 (2)
Thrombosis (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LMTM 100-300 mg/Day (N=896)
Anaemia (Blood and lymphatic system disorders) | 43 (45)
Diarrhoea (Gastrointestinal disorders) | 123 (174)
Nausea (Gastrointestinal disorders) | 44 (56)
Constipation (Gastrointestinal disorders) | 18 (19)
Vomiting (Gastrointestinal disorders) | 36 (40)
Fatigue (General disorders) | 20 (23)
Urinary tract infection (Infections and infestations) | 49 (72)
Lower respiratory tract infection (Infections and infestations) | 18 (21)
Nasopharyngitis (Infections and infestations) | 27 (31)
Upper respiratory tract infection (Infections and infestations) | 27 (34)
Fall (Injury, poisoning and procedural complications) | 62 (79)
Blood creatine phosphokinase increased (Investigations) | 21 (21)
Creatinine renal clearance decreased (Investigations) | 33 (37)
Haemoglobin decreased (Investigations) | 40 (44)
Weight decreased (Investigations) | 30 (31)
Arthralgia (Musculoskeletal and connective tissue disorders) | 27 (34)
Back pain (Musculoskeletal and connective tissue disorders) | 18 (21)
Dizziness (Nervous system disorders) | 23 (31)
Headache (Nervous system disorders) | 29 (33)
Agitation (Psychiatric disorders) | 46 (59)
Anxiety (Psychiatric disorders) | 32 (35)
Confusional state (Psychiatric disorders) | 34 (39)
Depression (Psychiatric disorders) | 21 (21)
Insomnia (Psychiatric disorders) | 19 (21)
Pollakiuria (Renal and urinary disorders) | 55 (58)
Urinary incontinence (Renal and urinary disorders) | 60 (67)
Dysuria (Renal and urinary disorders) | 39 (45)
Micturition urgency (Renal and urinary disorders) | 29 (30)
Cough (Respiratory, thoracic and mediastinal disorders) | 24 (24)
Hypertension (Vascular disorders) | 20 (20)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2016-03-24): https://cdn.clinicaltrials.gov/large-docs/68/NCT02245568/Prot_000.pdf
  • Statistical Analysis Plan (2017-03-30): https://cdn.clinicaltrials.gov/large-docs/68/NCT02245568/SAP_001.pdf